CLINICAL TRIAL: NCT05521581
Title: THE EFFECT OF AFTER CAESARIAN SECTION HAND MASSAGE ON PAIN, COMFORT LEVEL AND GAS OUTPUT TIME
Brief Title: Effects Of Hand Massage After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sinem Dügeroğlu, Principal İnvestigator, Selcuk University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukU SDugeroglu071
Record Dates: First submitted 2022-08-20; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Primiparous Mothers Who Gave Birth by Cesarean Section
Keywords: hand massage; cesarean delivery; ache; comfort; gas outlet; midwife
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
  Women who had cesarean section in the institution were evaluated in terms of sample.
  They were divided into two groups as criteria and random sampling. be an order obtained a random number table, capable of random sampling automatically by means of programs on websites by specifying a number. samples. Selection of intervention and control groups determined by tossing a coin. The sample number was determined as 83 women who had a total of 166 cesarean section in each of the intervention and control groups. Considering the data losses, 10% more was calculated and it was planned to conduct the research with a total of 182 women (91 women in the intervention group, 91 women in the control group).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Hand massage will be applied to primiparous mothers who gave birth by cesarean section
  Interventions: Other: Hand massage
- control (No Intervention): Routine care will be given to mothers who have given cesarean section and hand massage will not be applied.

INTERVENTIONS:
Other: Hand massage — Hand massage will be applied to primiparous mothers who gave birth by cesarean section and its effect on pain, comfort and gas release times will be evaluated.
  Arms: intervention

SUMMARY:
H1-1 Hypothesis: Hand massage applied after cesarean delivery has an effect on reducing the level of pain in the cesarean section incision area of women.

H1-2 Hypothesis: Hand massage applied after cesarean delivery has an effect on increasing the comfort scale score of women.

H1-3 Hypothesis: Hand massage applied after cesarean delivery has an effect on reducing the time of gas production in women.

ELIGIBILITY:
Inclusion Criteria:

Having primiparous pregnancy,

* 18 years old and over,
* Able to speak Turkish and express himself in Turkish,
* Does not have any disability (such as vision, hearing)
* Having completed the 6th hour after cesarean delivery, hospitalized in the gynecology service,
* Having undergone cesarean section with spinal anesthesia,
* Having no findings such as wounds, nerve problems, history of surgery or amputation on their hands,
* Single pregnancy,
* Women who are open to communication and who are mentally and physically healty

Exclusion Criteria:

Not accepting to work,

* Having a gas outlet before starting the application,
* Presence of findings such as wounds on hands, nerve problems, history of surgery or amputation,
* Having postpartum hemorrhage,
* With uterine subinvolution,
* Having a cesarean section with another type of anesthesia other than spinal anesthesia (such as general, epidural combined)
* Having twin babies,
* Having a premature baby (the baby needs more attention and care)
* Women whose babies are hospitalized in the neonatal intensive care unit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — primiparous women who had a cesarean section
Enrollment: 182 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
inclusion of women in the study and filling out the introductory information form | maximum one hour
  Women are included in the study by filling out the introductory information form. The information obtained will be recorded in the SPSS 20.0 package program.
ensuring the randomization of the women included in the study into the intervention and control groups | Five min
  Distributions are made to women included in the study and to control and intervention groups.
practicing and observing hand massage | an average of 12-13 hours
  Mothers assigned to the intervention group receive 2 sessions of hand massage. The first session is applied at the 6th hour after the cesarean section, and the second session is applied at the 12th hour after the cesarean section.
  Routine care is applied to the control group and hand massage is not applied.
assessment of pain | five min
  Women in the intervention and control groups are assessed for pain with the Visual Analog Scale (VAS).
comfort assessment | ten min
  Women in the intervention and control groups will be evaluated with the Postpartum Comfort Scale.
Evaluation of gas exit time | five min
  The effectiveness of hand massage will be evaluated by looking at the time between cesarean section hours and gas release times of women in the intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinem Dügeroğlu, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No